CLINICAL TRIAL: NCT06033287
Title: Observational Real-World Study on the Efficacy, Safety, and Biomarker Exploration of CDK4/6 Inhibitors Combined With Endocrine Therapy and Subsequent Treatment in HR+/HER2- Metastatic Breast Cancer.
Brief Title: Real-World Study on CDK4/6 Inhibitors Combined With Endocrine Therapy and Subsequent Treatment in HR+/HER2- MBC.
Status: Recruiting | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYJJ-2023-095
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer; Endocrine Therapy; CDK4/6 Inhibitors; Subsequent Treatment
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CDK4/6 inhibitors treatment: All HR+/HER2- metastatic breast cancer patients using CDK4/6 inhibitors
  Interventions: Drug: Different treatment regimens following progression on CDK4/6 inhibitors.

INTERVENTIONS:
Drug: Different treatment regimens following progression on CDK4/6 inhibitors. — This study is a single-arm, non-interventional study that evaluates the efficacy and safety of the first-line treatment regimen, which includes CDK4/6 inhibitors combined with endocrine therapy. After disease progression on first-line treatment, the second-line systemic treatment regimen (including but not limited to switching to another CDK4/6 inhibitor combined with endocrine therapy, other types of endocrine therapy, chemotherapy, targeted therapy, etc.) will be evaluated.

SUMMARY:
Exploring the Efficacy and Safety of Different Systemic Treatment Regimens after CDK4/6i Progression in the Real World has significant implications. This study is an observational, real-world study. It plans to include over 300 eligible HR+/HER2- metastatic breast cancer patients who are currently receiving or planning to receive endocrine therapy regimens containing CDK4/6 inhibitors. This study is a single-arm, non-interventional study that evaluates the efficacy and safety of the first-line treatment regimen, which includes CDK4/6 inhibitors combined with endocrine therapy, based on clinical guideline consensus. After disease progression on first-line treatment, the second-line systemic treatment regimen (including but not limited to switching to another CDK4/6 inhibitor combined with endocrine therapy, other types of endocrine therapy, chemotherapy, targeted therapy, etc.) will be chosen by the physician, and the efficacy and safety of subsequent treatment will be evaluated. Additionally, peripheral blood ctDNA testing will be used to assess changes in baseline and progression-related biomarkers, including ESR1, PI3KCA, FGFR1, PTEN, among some patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria:

  * Age ≥ 18 years, postmenopausal or pre/perimenopausal females, or male patients. Female patients must meet one of the following criteria:

    1. Prior bilateral oophorectomy or age ≥ 60 years.
    2. Age < 60 with natural postmenopausal status (defined as spontaneous cessation of regular menstruation for at least 12 consecutive months without any other pathological or physiological reasons), and estradiol (E2) and follicle-stimulating hormone (FSH) levels consistent with postmenopausal range.
    3. Pre/perimenopausal females may also be eligible but must be willing to receive LHRH agonist during the study.
  * Pathologically confirmed HR-positive male/female breast cancer patients with evidence of localized recurrence or metastasis, who are not suitable for curative surgery or radiation therapy:

ER-positive and/or PR-positive defined as the proportion of positively stained tumor cells ≥ 1% of all tumor cells (as confirmed by the investigators at the participating center).

* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* No prior systemic treatment or currently receiving CDK4/6 inhibitors as first-line treatment for advanced disease.
* Reproductive-age females must have a negative serum pregnancy test within 28 days before enrollment and male/female patients must be willing to use a medically approved highly effective contraceptive measure during the study period and up to 1 year after the last dose of investigational drug.
* Non-pregnant or non-lactating females.
* Not concurrently participating in any other ongoing study.
* Patient or legally authorized representative has provided informed consent and is willing and able to comply with the planned visits, study treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

* 1. Any evidence of severe or uncontrolled systemic illnesses, including uncontrolled hypertension, active bleeding disorders, active infections including hepatitis B, hepatitis C, and human immunodeficiency virus, or severely impaired bone marrow reserve or organ function, including liver and kidney impairment, which, in the investigator's opinion, would greatly alter the risk/benefit balance.
* Patient has not yet recovered from any CTCAE grade ≥ 3 toxicity related to prior treatment at the start of CDK4/6 inhibitor therapy.
* Known history of allergy to CDK4/6 inhibitors, excipients, or drugs with a similar chemical structure or class as CDK4/6 inhibitors.
* Patients deemed unsuitable for enrollment by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HR+/HER2- metastatic breast cancer patients who are currently receiving or planning to receive endocrine therapy regimens containing CDK4/6 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  The survival time from the date of randomization to the date of the first documented progression or date of death, whichever came first, assessed up to 36 months

SECONDARY OUTCOMES:
Objective Response Rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 36 months
  It is a statistical measure used in clinical trials to evaluate the effectiveness of a treatment by assessing the proportion of patients who achieve either a partial or complete objective response to the treatment.

OTHER OUTCOMES:
Overall survival | The time from randomization to death from any cause, whichever came first, assessed up to 36 months
  The time from randomization to death from any cause
Adverse Events | Primary Outcome Measure: 1.Progression-Free Survival The survival time from the date of randomization to the date of the first documented progression or date of death, whichever came first, assessed up to 60 months [Time Frame: From date of randomizatio
  All adverse events [including adverse events (AE / SAE) and ADR (adverse drug reactions)] will be collected when known. The classification of adverse reactions shall refer to CTCAE5.0 in case of adverse events / reactions. In case of serious adverse events, the investigators must immediately take necessary treatment measures to protect the safety of subjects. All adverse events / reactions should be tracked and observed. If the adverse events have not recovered, the investigator shall continue to give necessary treatment, report and record, and deal with special cases according to the management opinions of relevant departments.

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No